CLINICAL TRIAL: NCT04753203
Title: A Phase lb/ll, Open Label, Single Arm Study to Assess Efficacy and Safety of Alpelisib and Capecitabine in Patients With PIK3CA Mutant Metastatic Colorectal Cancer Who Failed Two Prior Standard Chemotherapies
Brief Title: Alpelisib and Capecitabine in Patients With PIK3CA Mutant mCRC Patients
Acronym: ALCAP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, SoohyeonLee, Assistant Professor, Korean Cancer Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2020-2011-003
Record Dates: First submitted 2021-02-04; First posted 2021-02-15 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Colorectal Cancer; PIK3CA Gene Mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Alpelisib

STUDY DESIGN:
Intervention Model Description: A phase lb/ll, open label, single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A single arm study with Alpelisib plus Capecitabine (Experimental): A phase lb/ll, open label, single arm study with Alpelisib plus Capecitabine in patients with PIK3CA mutant metastatic colorectal cancer
  Interventions: Drug: Alpelisib plus Capecitabine combination

INTERVENTIONS:
Drug: Alpelisib plus Capecitabine combination — Adding Alpelisib to Capecitabine as a salvage regimen in mCRC with PIK3CA mutation

SUMMARY:
The investigator assesses the efficacy and safety of alpelisib and capecitabine in patients with PIK3CA mutant metastatic colorectal cancer who failed two prior standard chemotherapies.

DETAILED DESCRIPTION:
Phase lb To determine maximal tolerated dose (MTD) and recommended phase ll dose (RP2D) of alpelisib in combination with capecitabine regardless of PIK3CA mutation of any solid tumors

Phase ll To investigate the progression-free survival (PFS)

Conduct the exploratory biomarker analysis for efficacy and resistance of alpelisib plus capecitabine combination (using collected clinical samples)

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed the Informed Consent Form (ICF) prior to any screening procedures being performed
2. Age ≥ 19 years old of male and female
3. At each phase of the trial, subjects who meet the following requirements in each phase will be enrolled.

   Phase Ib: Subjects with a histologically-confirmed, advanced/recurrent solid tumor who have progressed on standard therapy or whose disease does not have established standard therapy and not limited to PIK3CA mutation Phase II: Subjects with histologically confirmed, PIK3CA mutated, metastatic colorectal cancer that have progressed after treatment with two prior standard chemotherapeutic agents with targeted agents such as cetuximab, bevacizumab, aflibercept (Tissue samples of colorectal cancer patients must contain just PIK3CA gene alterations. e.g. single nucleotide variants, small indels, amplifications, structural variation etc. using targeted panel sequencing.)
4. Patient has evaluable disease as per RECIST 1.1. (Measurable lesions are not mandatory for study inclusion.)
5. ECOG performance status 0-1
6. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Hemoglobin ≥ 9.0 g/dL
   * Platelet ≥ 100 x 109/L
   * Serum creatinine ≤ ULN (upper limit of normal) or serum creatinine clearance > 50 mL/min
   * Total bilirubin: ≤ 1.5 × ULN Subjects with a bile duct obstruction will be eligible if they meet the criteria after appropriate bile drainage; Patients with Gilbert syndrome should also be included after confirming that the total bilirubin level is ≤ 1.5 x ULN in a follow-up screening test.
   * INR ≤1.5
   * Potassium within normal limits, or corrected with supplements
   * Fasting Serum amylase ≤ 2 × ULN
   * Fasting Serum lipase ≤ ULN

   Phase Ib: Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 3 x ULN (regardless of liver metastases) Phase II: AST and ALT ≤ 3 x ULN if liver metastases are absent, or AST and ALT ≤ 5 x ULN if liver metastases are present.
7. Adequate cardiac function: QTc ≤480 msec; if QTc exceeds 480 msec, subjects can be enrolled if the average QTc value is less than 480 msec by measuring 3 times consecutively in total.
8. The subject is able to swallow and retain oral medication
9. Serum β-HCG test negative within 14 days before the first administration of the study treatment (women of childbearing potential only).
10. Requirement for contraception must be observed by the subject.
11. Life expectancy of at least 3 months

Exclusion Criteria:

1. Patient has received previous treatment with a PI3K or AKT inhibitor. (Note prior mTOR inhibitor treatment is allowed.)
2. Patient has received previous capecitabine in metastatic setting.
3. Patient has a known or suspicious hypersensitivity to capecitabine or other products containing fluorouracil.
4. Any cytotoxic chemotherapy from a previous treatment regimen within 14 days. If the subject received an investigational drug from another clinical trial, the subject can be enrolled after 2 weeks of last administration and more than 5 x half-life of the investigational drug. If monoclonal antibody therapy was given, the subject can be enrolled after four weeks after the last does.
5. Active central nervous system (CNS) lesions (i.e., those with radiologically unstable or symptomatic brain lesions). For those who receive radiation or surgical treatment, the subject can be enrolled if the subject is maintained without steroid therapy and the evidence of CNS disease progression for more than 4 weeks. However, patients with leptomeningeal metastases are excluded.
6. Patient has currently documented pneumonitis/interstitial lung disease
7. Patient has not recovered to ≤ grade 1 (except alopecia) from related adverse effects of any prior anticancer therapy
8. Radiotherapy with a wide field (more than 30% of the bone marrow) of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment.
9. Patient who has undergone major surgery ≤ 4 weeks prior to starting study treatment or who has not recovered from adverse effects of such procedure.
10. Patient has a clinically significant cardiac disease or impaired cardiac function, such as:

    * Acute coronary syndrome within the 6 months prior to the initiation of study drug (including myocardial infarction or unstable angina, Coronary Artery Bypass Graft surgery, percutaneous coronary intervention and stenting)
    * Heart failure ≥ grade 2 by New York Heart Association (NYHA) functional classification or that requires treatment
    * Ejection fraction (EF) <50% on multi-gated acquisition (MUGA) scan or echocardiography examination. MUGA scan or echocardiography is not required as a screening test if there is no current suspicious symptom and past history of heart failure.
    * Persistent uncontrolled hypertension as defined by: systolic >160 mmHg or diastolic >100 mmHg with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.
    * Current or past history of clinically significant cardiac arrhythmia, atrial fibrillation, and/or conduction abnormality (e.g. congenital long QT syndrome, complete AV block)
    * On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or corrected QT (QTcF) >450 msec for males and >460 msec for females (using Fridericia's correction). All as determined by screening ECG (mean of triplicate ECGs).
    * Any risk factors that prolong QTc or increase the probability of arrhythmia, including medication (e.g. heart failure, hypokalemia, congenital long QT syndrome, history of Torsades de Pointes)
11. If the subject was diagnosed with diabetes (irrespective of treatment or symptom) or if the subject has impaired glucose tolerance (with blood glucose of 140-199 mg/dL after 2 hour oral glucose tolerance test (75g)), previous history of gestational diabetes, or steroid-induced diabetes.
12. Patients with impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. untreated peptic ulcer disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or wide small bowel resection).
13. History of acute pancreatitis within 1 year of screening or past medical history of chronic pancreatitis
14. Patient has a known positive serology for human immunodeficiency virus (HIV), active Hepatitis B, and/or active Hepatitis C infection. Hepatitis B carriers may be enrolled if prophylactic use of an antiviral agent with minimal interaction with CYP3A4 is administered to inhibit HBV activation (e.g., entecavir, adefovir)
15. Concomitant medication of strong or moderate inducers or inhibitors of CYP3A4 before the first dose of study treatment (In this case, if the drug is stopped for more than 1 week and changed to another drug that does not affect CYP3A4, then the subject can be enrolled.)
16. Inhibitors of BCRP
17. Subjects with unresolved osteonecrosis of the jaw
18. Subject has a history of severe cutaneous reactions like Stevens-Johnson-Syndrome (SJS), Erythema Multiforme (EM), Toxic Epidermal Necrolysis (TEN), or Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS).
19. History of other primary cancer. Exceptions are as follows:

    - Adequately treated non-melanoma skin cancer (basal cell or squamous cell carcinoma), curatively treated in situ cancer of the cervix or stage I bladder cancer, completely resected thyroid cancer without distant metastasis in which all treatment has been completed (Appropriate wound healing is required prior to clinical trial enrollment)
20. History of allogeneic bone marrow transplantation or organ transplantation
21. As judged by the Investigator, all other symptoms and associated disease for which the investigator determined that participation in this study is contraindicated (e.g. Infection/inflammation; severe liver dysfunction; bilateral diffuse interstitial lung disease; uncontrolled renal disease; unstable heart and lung disease; hemorrhagic disease; intestinal obstruction; unable to swallow oral pills; social and psychological problems, etc.)
22. Medical, psychiatric, cognitive, or other conditions that may interfere with the ability of the subject to understand the subject information, provide the informed consent, follow the protocol process, or complete the clinical trial

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-02-28 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerable dose | up to 6 month
  Maxiaml Tolerable Dose and Recommended Phase 2 Dose of combination Maximal tolerable dose and random phase 2 dose confirmation in Alpelisib with Capecitabine in phase 1b
Progression Free Survival | up to 3 years
  Progression Free Survival with RP2D dose

SECONDARY OUTCOMES:
Dose limiting toxicity | Up to 6 month
  Dose limiting toxicity
Objective response rate | up to 3 years
  Objective response rate (by RECIST v1.1)
Overall survival | up to 4 years
  Overall survival
Time to response | up to 3 years
  Time to response
Duration of response | up to 3 years
  Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Soohyeon Lee, MD, Principal Investigator — Korea Cancer Study Group
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No